CLINICAL TRIAL: NCT05952531
Title: Characterizing Myositis With 68Ga-FAPI PET/CT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI in IIM
Record Dates: First submitted 2023-07-12; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Myositis; Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Myositis | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — Intravenous injection of one dosage of 111-185 MBq (3-5 mCi) 68Ga-FAPI. Tracer doses of 68Ga-FAPI will be used to image IIM lesions in skeletal muscle, heart, lung, skin and potential tumor by PET/CT.
  Other Names: 68Ga-fibroblast activating protein inhibitor

SUMMARY:
To evaluate the potential usefulness of 68Ga-FAPI PET/CT for the diagnosis and evaluation of systemic involvement in idiopathic inflammatory myopathies (IIM)/myositis, and compared the results with those of 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Inflammatory myopathies (IIM), collectively known as myositis, are heterogeneous systemic autoimmune disorders characterized by muscle inflammation, and frequently accompanied by extra-muscular manifestations that affect the skin, lung, and joints. Prevalence of underlying malignancy is high in patients with IIM.

68Ga-FAPI has been developed as tracers specific for fibroblast-activation protein (FAP), which is overexpressed in activated fibroblasts in various type of cancers and autoimmune diseases, such as rheumatoid arthritis, IgG4-related diseases and interstitial lung diseases.

Recently the investigators have published articles of the application of 68Ga-FAPI in IgG4-related disease and rheumatoid arthritis, which showed it was more sensitive than FDG in detecting a certain type of inflammation, and the potential utility of FAP-targeted PET/CT imaging for disease assessment in myositis have been reported in a case recently.

Thus, this prospective study is going to investigate utility of 68Ga-FAPI PET/CT in diagnosis, disease assessment including skeletal muscle involvement, cardiac involvement, interstitial lung diseases and potential underlying cancer screening, response to treatment and prognosis, compared with 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of myositis according to American College of Rheumatology/European League Against Rheumatism 2017 (ACR/EULAR 2017) criteria
2. Adult men or women 18 and ≤ 75 years of age at the time of signing the informed consent (ICF).
3. Participants who were able to provide informed consent (signed by participant or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.
4. 68Ga-FAPI and 18F-FDG PET/CT were performed within two weeks.

Exclusion Criteria:

1. Pregnancy;
2. Breastfeeding;
3. known allergy against FAPI;
4. any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
To define the distribution pattern of 68Ga-FAPI in patients with IIM | 60 minutes following injection
  To quantify 68Ga-FAPI positron emission tomography (PET) tracer biodistribution in diseased tissue including muscle, heart, lung and normal background organs. 68Ga-FAPI positron emission tomography (PET) tracer biodistribution will be assessed by semi-quantitative analysis (unit/metrics = standardized uptake values (SUV)).

SECONDARY OUTCOMES:
Correlation between uptake of 68GA-FAPI and other parameters associated with disease activity | 30 days
  The Standardized uptake value (SUV) of 68Ga-FAPI was calculated and analyzing the correlation between pathological results and parameters associated with disease activity.
68Ga-FAPI and disease progression | Up to 2 years
  To evaluate whether the 68Ga-FAPI biodistribution in the diseased tissues can be associated with disease progression under therapies.
Therapy response | Up to 2 years
  To evaluate whether the change of 68Ga-FAPI uptake in diseased tissue can be associated with disease activity after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Guixiu Shi, PhD, Study Director — The First Affiliated Hospital of Xiamen University
Locations (1):
- The first affiliated hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No